CLINICAL TRIAL: NCT07177235
Title: Early Ketamine Plus Midazolam Versus Ketamine Plus Midazolam for the Treatment of Refractory Status Epilepticus
Brief Title: Ketamine for the Treatment of Refractory Status Epilepticus
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Syed Omar Shah, Associate Professor, Neurology and Neurological Surgery, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2025-0404
Record Dates: First submitted 2025-09-03; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Refractory Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Ketamine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early ketamine (Active Comparator): Initiation of ketamine infusion simultaneously with midazolam infusion as the third-line anesthetic treatment
  Interventions: Drug: Ketamine; Drug: Midazolam
- Late ketamine (Active Comparator): Initiation of ketamine infusion only after midazolam infusion has been started
  Interventions: Drug: Ketamine; Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Timing of ketamine initiation will differ between groups (early versus late ketamine)
Drug: Midazolam — Midazolam infusion will be initiated at the same time in both groups

SUMMARY:
This pilot feasibility study aims to examine how the timing of ketamine introduction as a third-line anti-seizure medication infusion relates to seizure cessation in patients with refractory status epilepticus (RSE).

DETAILED DESCRIPTION:
Patients admitted to the Jefferson Neurological Intensive Care Unit with seizures or status epilepticus will be screened for eligibility. Surrogate consent will be obtained from the participants legally authorized representative (LAR) by study personnel for eligible patients using remote e-consent process via RedCap. Participants will be randomized 1:1 to receive either early intravenous ketamine plus midazolam infusion or the current institutional protocol of midazolam followed by late ketamine infusion (Fernandez et al., 2018). Continuous video EEG monitoring will guide medication titration, increasing doses every 20 minutes for ongoing seizure activity. The primary goal of this study is to examine the feasibility of the protocol and obtain estimates of the timing of seizure cessation. The primary outcome is time to seizure cessation, defined as the time from initiation of anesthetic infusion (midazolam or midazolam plus ketamine) to the time of last electrographic seizure. The investigators will also collect preliminary data on other clinical measures that would serve as secondary outcomes for future trials. These clinical measures include progression to super refractory status epilepticus, intensive care unit and hospital length of stay, duration of mechanical ventilation, and functional outcomes assessed by the modified Rankin Scale at discharge, 3 months, and 6 months. This study does not evaluate ketamine as a novel therapy but rather assesses a minor modification in the timing of ketamine administration to optimize seizure control.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older
2. Patients with refractory status epilepticus unresponsive to appropriately dosed first line agents administered intravenous or intraosseous and one second line agent

   1. First line agents: lorazepam, midazolam, or diazepam
   2. Second line agents: phenytoin (20 mg/kg), valproate (40 mg/kg), levetiracetam (60 mg/kg), lacosamide (400 mg)
3. All etiologies of status epilepticus will be included

Exclusion Criteria:

1. Exclusively psychogenic non epileptic seizures
2. Pregnant individuals
3. Incarcerated individuals
4. Patients with hypersensitivity to ketamine or any component of the formulation
5. Conditions in which an increase in blood pressure would be hazardous
6. Focal motor status epilepticus
7. Status epilepticus lasting > 24 hours prior to enrollment (SRSE)
8. Patients with EEG in the ictal-interictal continuum (IIC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Time to seizure cessation | 72 hours
  Time from initiation of anesthetic infusion (midazolam or midazolam plus ketamine) to the time of last electrographic seizure

CONTACTS AND LOCATIONS:
Overall Officials: Syed O Shah, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Background] Bruno A, Akinwuntan AE, Lin C, Close B, Davis K, Baute V, Aryal T, Brooks D, Hess DC, Switzer JA, Nichols FT. Simplified modified rankin scale questionnaire: reproducibility over the telephone and validation with quality of life. Stroke. 2011 Aug;42(8):2276-9. doi: 10.1161/STROKEAHA.111.613273. Epub 2011 Jun 16. PMID 21680905
- [Background] Golub D, Yanai A, Darzi K, Papadopoulos J, Kaufman B. Potential consequences of high-dose infusion of ketamine for refractory status epilepticus: case reports and systematic literature review. Anaesth Intensive Care. 2018 Sep;46(5):516-528. doi: 10.1177/0310057X1804600514. PMID 30189827
- [Background] Janssen PM, Visser NA, Dorhout Mees SM, Klijn CJ, Algra A, Rinkel GJ. Comparison of telephone and face-to-face assessment of the modified Rankin Scale. Cerebrovasc Dis. 2010 Jan;29(2):137-9. doi: 10.1159/000262309. Epub 2009 Dec 1. PMID 19955737
- [Background] Legriel S, Oddo M, Brophy GM. What's new in refractory status epilepticus? Intensive Care Med. 2017 Apr;43(4):543-546. doi: 10.1007/s00134-016-4501-6. Epub 2016 Aug 20. No abstract available. PMID 27544138
- [Background] Trinka E, Cock H, Hesdorffer D, Rossetti AO, Scheffer IE, Shinnar S, Shorvon S, Lowenstein DH. A definition and classification of status epilepticus--Report of the ILAE Task Force on Classification of Status Epilepticus. Epilepsia. 2015 Oct;56(10):1515-23. doi: 10.1111/epi.13121. Epub 2015 Sep 4. PMID 26336950
- [Background] Fletman EW, Cleymaet S, Salvatore A, Devlin K, Pickard A, Shah SO. Ketamine plus midazolam compared to midazolam infusion for the management of refractory status epilepticus. Clin Neurol Neurosurg. 2024 Nov;246:108592. doi: 10.1016/j.clineuro.2024.108592. Epub 2024 Oct 12. PMID 39418930